CLINICAL TRIAL: NCT01377285
Title: Renoprotection by Combining Pentoxifylline and Angiotensin Blockade in Chronic Kidney Disease
Brief Title: Renoprotection by Pentoxifylline and Angiotensin Receptor Blocker in Chronic Kidney Disease (CKD)
Acronym: CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other); Mackay Memorial Hospital (Other); Taipei Medical University Hospital (Other); Shin Kong Wu Ho-Su Memorial Hospital (Other); Cathay General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200809041M
Record Dates: First submitted 2010-06-08; First posted 2011-06-21 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Renal Failure
Keywords: chronic kidney disease; pentoxifylline; angiotensin receptor blockers(ARB)
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic | interventions — Angiotensin Receptor Antagonists; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARB & Pentoxifylline (Experimental): angiotensin receptor blockers(ARB)and Pentoxifylline 400mg tablet (If CKD3 1# BID(Bi in die=two times a day); CKD4 1# QD(quaque die=one time a day); CKD5(estimated Glomerular filtration rate,eGFR<15ml/min/1.73 m2) 1# QOD(Every other day).
  Interventions: Drug: ARB; Drug: Placebo (for Pentoxifylline)
- ARB & Placebo (Active Comparator): angiotensin receptor blockers(ARB) and Placebo tablet(If CKD3 1# BIDBi in die=two times a day); CKD4 1# QD(quaque die=one time a day); CKD5(estimated Glomerular filtration rate,eGFR<15ml/min/1.73 m2) 1# QOD(Every other day).
  Interventions: Drug: Pentoxifylline; Drug: Placebo (for Pentoxifylline)

INTERVENTIONS:
Drug: ARB — Angiotensin II receptor antagonists ,these medicines have names that end in "sartan".For examples:losartan,candesartan,irbesartan,olmesartan,telmisartan,valsartan
  Other Names: angiotensin receptor blockers(ARB)
  Arms: ARB & Pentoxifylline
Drug: Pentoxifylline — This medication is used to improve the symptoms of a certain blood flow problem in the legs/arms (intermittent claudication due to occlusive artery disease)
  Other Names: Trental
  Arms: ARB & Placebo
Drug: Placebo (for Pentoxifylline) — Sugar pill manufactured to mimic Pentoxifylline 400mg tablet
  Other Names: Placebo(non treatment)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled clinical trial to investigate the renoprotective efficacy of combined pentoxifylline (PTX) and angiotensin receptor blockers (valsartan), compared with placebo and valsartan in 700 patients with Chronic Kidney Disease (CKD) stages 3 and 4. The effect on cardiovascular comorbidity will also be observed. The observation period will be 3 years. The primary endpoints consists of doubling of serum creatinine, end stage renal disease (ESRD), and death from any cause. The secondary endpoints include changes of microalbuminuria or proteinuria, serum and urinary levels of TNF-a(tumor necrosis factor-alpha ), MCP-1(monocyte chemotactic protein), TGF-beta1(transforming growth factor ), collagens III (amino terminal peptide of procollagen III) and IV, and fibronectin, urinary N-acetyl-beta-glucosaminidase, as well as serum fibrinogen and high-sensitive CRP(C reactive protein), and development of heart failure, nonfatal myocardial infarction, and stroke or transient ischemic attack.

DETAILED DESCRIPTION:
This study is a multicenter placebo-controlled double-blind randomized clinical trial. The design scheme is depicted in Figure 1. (see below). At the time of screening, all pentoxifylline-naïve participants must have been receiving angiotensin receptor blockers(ARB) per day for no less than 8 weeks and have stable renal function with serum creatinine elevation < 25% in the preceding 8 weeks. For patients taking maximal dose of angiotensin receptor blockers(ARB) for more than 8 weeks, randomization will be started after recruitment. For patients taking submaximal, fixed dose of angiotensin receptor blockers(ARB)for ≥ 8 weeks, with good BP(blood pressure), i.e., ≤ 130/80 mmHg, randomization can also be started after recruitment. However, for patients taking submaximal dose of angiotensin receptor blockers(ARB) with suboptimal BP, i.e., >130/80 mmHg, patients can be recruited but will not be randomized until the dose of angiotensin receptor blockers(ARB) has been fixed for ≥ 8 weeks, or a maximal dose of angiotensin receptor blockers(ARB) has been administered for ≥ 8 weeks.The recruited CKD(Chronic kidney disease) patients will be randomized to receive pentoxifylline (400 mg once or twice a day) or placebo (one tablet once or twice a day). Patients with stage 3 CKD(estimated GFR,eGFR30-59.9ml/min/1.73 m2) will receive either pentoxifylline one tablet (400 mg) twice a day, or placebo one tablet twice a day.If the patients are still intolerant of the potential side effects, they may withdraw from the study voluntarily. Patients with stage 4 CKD(estimated Glomerular filtration rate,eGFR15-29ml/min/1.73 m2) will receive either pentoxifylline one tablet (400 mg) once per day, or placebo one tablet once per day. In patients who develop potential side effects (anorexia, epigastric distention, dizziness, and headache) to the test drug, they may withdraw from the study voluntarily. If patients have SBP(systolic blood pressure ) > 130 mmHg and/or DBP (diastolic blood pressure )> 80 mmHg, it is necessary to adjust the other antihypertensive drugs. However, the following medications are not allowed during the study: ACE(angiotensin-converting-enzyme) inhibitor; phosphodiesterase inhibitor (other than pentoxifylline); direct vasodilators (e.g., hydralazine and minoxidil), as they can blunt the decrease in proteinuria, and chronic immunosuppressive or non-steroidal anti-inflammatory drug (NSAID) therapy.

The randomization is done with the stratifications of CKD(Chronic kidney disease) stages and diabetic/non-diabetic status. CKD includes stage 3(estimated GFR,eGFR30-59.9ml/min/1.73 m2) and 4(estimated Glomerular filtration rate,eGFR15-29ml/min/1.73 m2). CKD stage 3 is further divided to 3A(estimated Glomerular filtration rate,eGFR45-59ml/min/1.73 m2) and 3B(estimated Glomerular filtration rate,eGFR30-44ml/min/1.73 m2) according to most recent guideline (NICE clinical guideline 73, Chronic kidney disease, September 2008) Two-arm random permuted block randomization with mixed block sizes 6, 8 and 10 will be implemented within each stratum. Double-blind measures will be enforced in each participating hospital. And, extra efforts will be made to avoid noncompliance, missing data, and loss to follow-up during the trial. Patient's renal function will be calculated by the Cockcroft-Gault and simplified MDRD(Modification of Diet in Renal Disease) formula. All blood and urine analyses will be performed by the Department of Laboratory Medicine, NTUH(National Taiwan University Hospital). Serum and urine samples are collected before and annually after randomization, and the specimens are allocated and stored at -70°C. Profibrotic or inflammatory markers such as serum and urinary levels of TNF-alpha, MCP-1, TGF-beta1, collagens III(amino-terminal propeptide of type III procollagen) and IV, and fibronectin, urinary NAG, as well as serum fibrinogen and high-sensitive CRP will be measured by using commercially available kits. Genetic polymorphism of MCP-1 and fractalkine receptor will also be analyzed to evaluate their association with renal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic and non-diabetic men and women between 20 and 80 years of age who have been diagnosed as CKD stage 3 to 4. The diabetic patients must be type II diabetes mellitus (DM) having overt proteinuria or microalbuminuria twice within the preceding 6 months with a clinical exclusion of non-diabetic kidney diseases. Non-diabetic patients may or may not have overt proteinuria; for proteinuric non-diabetic patients, the proteinuria must be present on two occasions within the preceding 6 months.
* Renal replacement therapy is not expected within the forthcoming 12 months.
* Currently under angiotensin receptor blockers(ARB) therapy for at least 8 weeks, with systolic blood pressure<150 mmHg, diastolic blood pressure <90 mmHg
* Renal function has been stable for at least 8 weeks (fluctuation<25% of baseline) at the time of screening

Exclusion Criteria:

* Type I DM patients
* Patients with history of allergy to pentoxifylline or methylxanthine derivatives (such as caffeine, theophylline)or those who have been taking pentoxifylline or dipyridamole as a treatment for chronic disease in the preceding 3 months at screening.
* Patients have been taking ACE inhibitors, renin inhibitors (eg. Rasilez); and direct vasodilators (e.g., hydralazine and minoxidil) at the time of screening
* Females in nursing or pregnancy, or preparing for pregnancy within the next three years.
* Obstructive uropathy.
* Active gastrointestinal bleeding Active peptic ulcer, patients with active bleeding or bleeding tendency and patients under antiplatelet or anticoagulant therapy,except for aspirin 100 mg, clopidogrel 75 mg.
* Unable to stop chronic immunosuppressive therapy or NSAID; or current use of phosphodiesterase inhibitors other than pentoxifylline (eg., dipyridamole)
* Congestive heart failure of functional class III or IV.
* Unstable angina, myocardial infarction, coronary artery bypass graft surgery, or percutaneous coronary intervention, within the past 3 months prior to signing for informed consent.
* Cerebral vascular diseases within the past 3 months prior to signing for informed consent.
* Retinal hemorrhage within the past 3 months prior to signing for informed consent.
* Known or suspected secondary hypertension (e.g., primary aldosteronism, renovascular hypertension, and pheochromocytoma).
* Poor glycemic control (HbA1c>8.5%)
* Liver cirrhosis or hepatic dysfunction as defined by abnormal liver function test
* Biliary obstructive disorders (e.g., cholestasis).
* Active malignancy or infectious diseases.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2010-06; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
doubling of serum creatinine, ESRD, and death from any cause | 3 years

SECONDARY OUTCOMES:
changes of microalbuminuria or proteinuria, and development of heart failure, nonfatal myocardial infarction, and stroke or transient ischemic attack. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Ming Chen, M.D.; PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
if the subject have serious adverse event and Data Monitoring Committee decide need to make individual participant data,study team will provide data.